CLINICAL TRIAL: NCT06339008
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Lebrikizumab/ LY3650150 in Adult Participants With Perennial Allergic Rhinitis
Brief Title: A Study of Lebrikizumab in Adult Participants With Perennial Allergic Rhinitis (PREPARED-1)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18789; J2T-MC-KGBT (Other: Eli Lilly and Company); 2023-508817-18-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Perennial Allergic Rhinitis (PAR)
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lebrikizumab every 2 weeks (Q2W)/ every 4 weeks (Q4W) (Experimental): Lebrikizumab will be given as a subcutaneous (SC) injection. Participants will receive background therapy with intranasal corticosteroids (INCS).
  Interventions: Drug: LY3650150; Drug: Standard therapy for INCS
- Lebrikizumab Q2W/every 8 weeks (Q8W) (Experimental): Lebrikizumab will be given as an SC injection. Participants will receive background therapy with INCS.
  Interventions: Drug: LY3650150; Drug: Standard therapy for INCS
- Placebo Q2W/Q4W (Placebo Comparator): Placebo matching Lebrikizumab will be given as an SC injection. Participants will receive background therapy with INCS.
  Interventions: Drug: Placebo; Drug: Standard therapy for INCS

INTERVENTIONS:
Drug: LY3650150 — Administered SC
  Arms: Lebrikizumab Q2W/every 8 weeks (Q8W); Lebrikizumab every 2 weeks (Q2W)/ every 4 weeks (Q4W)
Drug: Placebo — Administered SC
  Arms: Placebo Q2W/Q4W
Drug: Standard therapy for INCS — Administered as intranasal spray

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of lebrikizumab in adult participants with perennial allergic rhinitis.

Participants can expect study participation to last up to 29.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed perennial allergic rhinitis (PAR).
* Has a positive skin prick test (SPT) with indoor allergens and/or positive serum antigen-specific immunoglobulin E (IgE) for indoor allergens ≥0.70 kU/L, utilizing a validated assay (central laboratory).
* The participant must have clinical symptoms at study entry associated with positive perennial allergen as tested by the SPT or a positive serum antigen-specific IgE test.
* A participant who has a known history of dermatographism or identified during the SPT may participate in this study with a positive serum antigen-specific IgE test.
* Participants who have concomitant asthma must be stable in the 3 months prior to screening using permitted regular asthma treatment.

Exclusion Criteria:

* Have received a dose of lebrikizumab.
* Is currently on AIT subcutaneous immunotherapy or sublingual immunotherapy. However, individuals who discontinued subcutaneous or sublingual immunotherapy for ≥3 years prior to randomization are eligible.
* Have received treatment with any rescue medication during the run-in period.
* Have received treatment with any biologic or systemic immunosuppressants, including Janus Kinase inhibitors (JAK) for inflammatory disease or autoimmune disease prior to the baseline visit:

  * Any current or prior use of biologics indicated for asthma or AD are prohibited.
  * B cell-depleting biologics, including rituximab, within 6 months.
  * Other biologics within 5 half-lives (if known) or 8 weeks, whichever is longer.
  * Systemic immunosuppressants, including JAK inhibitors, within 4 weeks prior to baseline.
* Have a history of seasonal worsening of AR and if the seasonal worsening is expected during the 4-week run-in period, the first 16 weeks after randomization, or during the last 8 weeks of the maintenance period.
* Anticipates significant changes in their daily environmental exposure.
* Has a known history of recurrent acute or chronic sinusitis.
* Female participant who is pregnant, breastfeeding or is planning to become pregnant or to breastfeed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline (CFBL) in Total Nasal Symptom Score (TNSS) at Week 16 | Baseline, Week 16
  Total nasal symptom score was a composite of 4 symptoms (rhinorrhea, nasal congestion, nasal itching and sneezing), each symptom was scored on a scale of 0 = none, 1 = mild, 2 = moderate, 3 = severe. The total score ranged from 0 to 12. The higher the score was, the more severe the symptoms were.

SECONDARY OUTCOMES:
Mean CFBL in Rhinoconjunctivitis Quality of Life Questionnaire Standardized Version [RQLQ(S)] Activities Domain at Week 16 | Baseline, Week 16
  The RQLQ includes 28 questions (completed between 10-15 min). Participants are asked to recall their experiences during the previous week and to respond to each question on a 7-point scale. The RQLQ score ranges from 0 to 6 (0 = no impairment, 6 = severe impairment).
Mean CFBL in RQLQ(S) Activities Domain at Week 56 | Baseline, Week 56
  The RQLQ includes 28 questions (completed between 10-15 min). Participants are asked to recall their experiences during the previous week and to respond to each question on a 7-point scale. The RQLQ score ranges from 0 to 6 (0 = no impairment, 6 = severe impairment)
Mean CFBL in RQLQ(S) Total Score at Week 16 | Baseline, Week 16
  The RQLQ includes 28 questions (completed between 10-15 min). Participants are asked to recall their experiences during the previous week and to respond to each question on a 7-point scale. The RQLQ score ranges from 0 to 6 (0 = no impairment, 6 = severe impairment).
Mean CFBL in RQLQ(S) Total Score at Week 56 | Baseline, Week 56
  The RQLQ includes 28 questions (completed between 10-15 min). Participants are asked to recall their experiences during the previous week and to respond to each question on a 7-point scale. The RQLQ score ranges from 0 to 6 (0 = no impairment, 6 = severe impairment).
Mean CFBL in TNSS at Week 4 | Baseline, Week 4
  Total nasal symptom score was a composite of 4 symptoms (rhinorrhea, nasal congestion, nasal itching and sneezing), each symptom was scored on a scale of 0 = none, 1 = mild, 2 = moderate, 3 = severe. The total score ranged from 0 to 12. The higher the score was, the more severe the symptoms were.
Mean CFBL in TNSS at Week 56 | Baseline, Week 56
  Total nasal symptom score was a composite of 4 symptoms (rhinorrhea, nasal congestion, nasal itching and sneezing), each symptom was scored on a scale of 0 = none, 1 = mild, 2 = moderate, 3 = severe. The total score ranged from 0 to 12. The higher the score was, the more severe the symptoms were.
Mean CFBL in Postnasal Drip Score at Week 16 | Baseline, Week 16
  Postnasal drip is mucus drainage down the throat, as part of their Allergic Rhinitis (AR), will be rated by participants using a 4-point scale, where 0 corresponds to no symptoms and 3 corresponds to severe symptoms. Study participants are asked to record the severity of their postnasal drip, at its worst, for the previous 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (74):
- United States (26):
  - Allergy and Asthma Specialists Medical Group, Huntington Beach, California
  - 310 Clinical Research, Inglewood, California
  - Allergy & Asthma Associates of Southern California dba. Southern California Research, Laguna Niguel, California
  - Allergy and Asthma, San Diego, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Allergy and Asthma Diagnostic Center, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Asthma Allergy Center of Chicago, River Forest, Illinois
  - Bluegrass Allergy Research, Lexington, Kentucky
  - Respiratory Medicine Research Institute of Michigan, PLC, Ypsilanti, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - University of Missouri Hospital, Columbia, Missouri
  - Allergy and Asthma Consultants, St Louis, Missouri
  - Asthma and Allergy Center, Bellevue, Nebraska
  - Circuit Clinical/Hudson-Essex Allergy, Belleville, New Jersey
  - Circuit Clinical/Mercer Allergy and Pulmonary Associates, Hamilton, New Jersey
  - Dr. Patrick Perin, Teaneck, New Jersey
  - Smith Allergy and Asthma, Horseheads, New York
  - Allergy Partners, Asheville, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Northwest Research Center, Portland, Oregon
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - AARA Research Center, Dallas, Texas
  - Kerrville Allergy and Asthma Associates, Kerrville, Texas
  - Allergy, Asthma & Sinus Center, Greenfield, Wisconsin
- Belgium (5):
  - Hôpital Erasme, Service Pharmacie, Brussels
  - Pneumocare, Erpent
  - UZ Gent, Ghent
  - UZ Leuven, Pharmacy, Leuven
  - Hôpital de la Citadelle, Liège
- China (17):
  - Internal Medicine Building, Beijing
  - Department of Nasal Allergy, Beijing
  - The Third Xiangya Hospital of Central South University, Changsha
  - GCP Pharmacy, Guangzhou
  - Zhejiang People's Hospital, Hangzhou
  - Jingzhou Central Hospital, Jingzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Tongji Hospital, Shanghai
  - Outpatient building, Wuhan
  - Outpatient Department, Union Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Northern Jiangsu People's Hospital, Yangzhou
  - Yangzhou University, Yangzhou
  - Zhongshan City People's Hospital, Zhongshan
- Germany (7):
  - Charité - Universitätsmedizin Berlin Klinik für Dermatologie, Berlin
  - Praxis für HNO und Allergologie, Dresden
  - Universitätsklinikum Carl Gustav Carus an der TU, Dresden
  - IKF Pneumologie, Frankfurt am Main
  - Siteworks - Zentrum für klinische Studien Heidelberg, Heidelberg
  - Universitätsklinik Marburg,Hals-, Nasen- und Ohrenklinik, Sektion Rhinologie und Allergologie, Marburg
  - Zentrum für Rhinologie und Allergologie, Weisbaden
- Poland (11):
  - Polimedica PTG Kielce, Kielce
  - Centrum Medyczne Promed ul. Olszańska 5G, Krakow
  - Malopolskie Centrum Alergologii, Krakow
  - gab. 114, ul. inż. pilota Wigury, Lodz
  - ETG Lublin, Lublin
  - Centrum Alergologii Teresa Hofman Sp z.o.o., Piła
  - EMED Centrum Usług Medycznych, Rzeszów
  - ClinMedica Research, Skierniewice
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp Z O.O., Tarnów
  - ETG Warszawa, Warsaw
  - ALL-MED - Specjalistyczna Opieka Medyczna, Wroclaw
- South Korea (8):
  - Inje University Haeundae Paik Hospital, Busan
  - B1F, Pharmacy department, Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kyunghee University Hospital at Gangdong, Seoul
  - Gangnam Severance Hospital 211, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Clinical trial Pharmacy, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement
URL: http://vivli.org/